CLINICAL TRIAL: NCT01832298
Title: Phase I Study of Simmitecan Hydrochloride for Injection in Patients With Advanced Solid Tumor：Tolerability and Pharmacokinetics
Brief Title: Study of Simmitecan Hydrochloride in the Treatment of Advanced Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Haihe Biopharma Co., Ltd. (Industry)
Collaborators: Shanghai Institute of Materia Medica, Chinese Academy of Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LP-101
Record Dates: First submitted 2013-04-08; First posted 2013-04-16 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-10

CONDITIONS: Advanced Solid Tumor
Keywords: Tolerability; Pharmacokinetics
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Simmitecan Hydrochloride for Injection (Experimental): Dissolving in 2ml water for injection, then transfering to 500 mL of 5% dextrose for i.v.90 minutes
  Interventions: Drug: Simmitecan Hydrochloride for Injection

INTERVENTIONS:
Drug: Simmitecan Hydrochloride for Injection — Either at 12.5 mg, 25 mg、50 mg、80 mg、120 mg、160 mg、200 mg

SUMMARY:
RATIONAL: Simmitecan is an anticancer ester prodrug, which involves activation to chimmitecan. Chimmitecan，a novel CPT derivative, exhibited potent antitumor activities both in vitro and in vivo by inhibiting topoisomerase I. Also exerted comparable effects on topoisomerase I compared with topotecan and SN38 and possessed improved anticancer potency and pharmacologic profiles, compared with the clinically available CPT analogues.

PURPOSE: to determine the maximum tolerated dose, the safety profile and pharmacokinetics of Simmitecan.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory to standard therapy or no standard therapy available.
* At least one measurable lesion.
* Age = 18~65 years.
* ECOG=0-1.
* Life expectancy ≥ 12 weeks.
* More than 4 weeks after operation, chemotherapy, radiotherapy, cytotoxic agents or tyrosine kinase inhibitors.
* Adequate organ function:

Haemoglobin ≥ 100 g/L, Absolute neutrophil count [ANC] ≥ 2×109/L,Platelets ≥ 100 × 109/L), Serum bilirubin ≤ 1.0×ULN, Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) < 1.5×ULN (If liver metastases, serum transaminase ≤ 2.5×ULN), Creatinine clearance ≥ 50 mL/min , LVEF ≤ 50%, QT interval (corrected by Fridericia): male < 450 ms, female < 470 ms

* Female: All subjects who are not surgically sterile or postmenopausal must agree and commit to the use of a reliable method of birth control for the duration of the study and for 6 months after the last dose of test article. Child bearing potential, a negative urine or serum pregnancy test result before initiating Famitinib. Male: All subjects who are not surgically sterile or postmenopausal must agree and commit to the use of a reliable method of birth control for the duration of the study and for 6 months after the last dose of test article.
* Signed and dated informed consent. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedure.

Exclusion Criteria:

* Less than 4 weeks from the last clinical trial.
* Known Spinal Cord compression or diseases of brain or pia mater by CT /MRI screening.
* Patients had ever severe diarrhea with prior therapy of camptothecin drugs.
* Concurrent severe or uncontrolled medical disease (serious infection, serious diabetes)
* Significant cardiovascular disease or condition including ≥ class II cardiac function (NYHA)
* Acute and chronic viral hepatitis. (If HBsAg +, HBV-DNA quantification ≤ LLN.)
* Pregnant, lactation period or men/women ready to birth.
* Psychiatric disorder or altered mental status.
* Evidence of significant medical illness that in the investigator's judgment will substantially increase the risk associated with the subject's participation in and completion of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2012-12; Primary Completion 2016-03 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) and maximum tolerated dose (MTD) | 2 weeks
  To evaluate the DLT and MTD in patients with advanced solid tumor

SECONDARY OUTCOMES:
Pharmacokinetic Assessment | 1-4 days
  To investigate pharmacokinetics of Simmitecan and Chimmitecan:AUC,Cmax,T1/2, CL/F.
Efficacy Assessments | 0-6 weeks
  Objective Response Rate (ORR), Disease Control Rate(DCR)
Pharmacodynamic Assessments | 0 days
  Evaluate the genotyping of UGT1A1*6 and UGT1A1*28.

CONTACTS AND LOCATIONS:
Overall Officials: Jinwan Wang, M.D., Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Aiping Zhou, M.D., Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Yong Xu, M.D., Principal Investigator — West China Hospital; Qingyuan Zhang, M.D., Principal Investigator — The Tumor Hospital Affiliated to Harbin Medical University
Locations (3):
- China (3):
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - The tumor hospital affiliated to Harbin medical university, Harbin, Heilongjiang
  - West China Hospital, Sichuan University, Chengdu, Sichuan